CLINICAL TRIAL: NCT04457570
Title: ONCOVID-AURA: Excess Risk of Morbi-mortality Due to COVID-19 in Patients With Cancer
Brief Title: Excess Risk of Morbi-mortality Due to COVID-19 in Patients With Cancer
Acronym: ONCOVID-AURA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0509
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: COVID, Cancer
MeSH Terms: conditions — Neoplasms | interventions — Mortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed patients: The "exposed patients" are patients with cancer that are hospitalized in one of the participating centers for a SARS-CoV-2 infection. A patient will be considered as an "exposed patient" if he/she had a surgical procedure or a medical treatment for cancer in the past 5 years preceding the SARS-CoV-2 infection.
  Interventions: Other: mortality
- control patients: The "control patients " are all of the patients without cancer that are hospitalized in one of the participating centers for a SARS-CoV-2 infection
  Interventions: Other: mortality

INTERVENTIONS:
Other: mortality — To measure the excess risk of mortality of patients with a history of cancer among patients hospitalized for a SARS-CoV-2 infection

SUMMARY:
Context:

Based on currently available data, most of national health authorities and consensus expert groups have written guidelines for the management of cancer patients in the context of COVID. However, the preparation of these guidelines was limited by the scarcity of solid epidemiological data. For example, the experts were uncomfortable to formulate precise guidelines on which anti-cancer treatment should be interrupted or replaced, on which patients, and how to adapt supportive drug prescriptions.

Objectives :

* To measure the excess risk of mortality and morbidity of patients with a history of cancer among patients hospitalized for a SARS-CoV-2 infection.
* To identify factors associated with the risk of death and morbidity among patients with cancer.

Methodology:

Retrospective inclusion of n=200 cancer patients hospitalized for COVID and n=400 matched (based on age, gender, and comorbidity) non-cancer patients hospitalized for COVID. Two analyses will be performed (after the inclusion of n=100 and n=200 patients with cancer). A logistic modeling of the odds ratio of death associated to the exposition factor (i.e. cancer) and adjusted for the matching parameters (age, gender, comorbidities) will be proposed.

We will then look for the factors (related to the patients, the cancer or the treatment) that modify the odds radio.

Expected results:

The data generated will help the medical and scientific community to evaluate the increasing risk of cancer patients infected by SARS-CoV-2 compared to the non-cancer population, to identify patients at higher risk of severe infection, but also the anticancer treatments associated with an increased risk of severe infections.

Impact:

These data will contribute to guide the future recommendations concerning cancer patient's care in the context of the COVID-19 pandemic. There is a real risk that the SARS-CoV epidemic, or other respiratory viruses epidemic, will become recurrent in the future. Thus, it is of crucial importance for now and for the future to know which are the major factors associated with severe infections

ELIGIBILITY:
Inclusion Criteria:

* EXPOSED PATIENTS:
* Age > 18 years old
* Patients with a confirmed diagnosis of solid or hematologic cancer
* Patients who received their last anticancer treatment (surgery, systemic treatments or other localized treatment) in the past 5 years before SARS-CoV-2 infection
* Positive laboratory test (RT-PCR) proving the SARS-CoV-2 infection
* Patients hospitalized in one of the participating centers because of the SARS-CoV-2 infection
* Patients who are not opposed in participating to the ONCOVID-AURA study

CONTROL PATIENTS:

* Age > 18 years old
* Patients who have no cancer (neither solid nor hematologic tumors) or patients who received their last anticancer treatments more than five years before the SARS-CoV-2 infection
* Positive laboratory test (RT-PCR) proving the SARS-CoV-2 infection
* Patients hospitalized in one of the participating centers because of the SARS-CoV-2 infection
* Patients who are not opposed in participating to the ONCOVID-AURA study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two categories of patients will be defined: the "exposed patients" are patients with cancer that are hospitalized in one of the participating centers for a SARS-CoV-2 infection. A patient will be considered as an "exposed patient" if he/she had a surgical procedure or a medical treatment for cancer in the past 5 years preceding the SARS-CoV-2 infection.
  The "control patients" are all of the patients without cancer that are hospitalized in one of the participating centers for a SARS-CoV-2 infection.
  In both cohorts, a positive laboratory test (RT-PCR) proving the SARS-CoV-2 infection will be mandatory.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
mortality for SARS-CoV-2 infection | 30 days
  mortality within 30 days after the hospitalization for the SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre de lutte contre le Cancer JEAN PERRIN, Clermont-Ferrand
  - Centre Hospitalier Uniersitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire de St Etienne, Saint-Etienne
  - Institut de Cancérologie de la Loire Lucien Neurwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: Undecided